CLINICAL TRIAL: NCT03653104
Title: Melodica Orchestra for Dyspnea: Safety and Feasibility Pilot
Acronym: MELODY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not initiate study intervention.
Sponsor: VA Quality Enhancement Research Intiative (Other)
Responsible Party: Principal Investigator, Dawn M. Bravata, Professor of Medicine & Adjunct Professor of Neurology, VA Quality Enhancement Research Intiative
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1802361245
Record Dates: First submitted 2018-08-21; First posted 2018-08-31 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2019-09

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease; Dyspnea; Breathlessness; Emphysema; Chronic Bronchitis
Keywords: Melodica; pursed lip breathing; breathing exercise; Music
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Intervention Model Description: This is a safety and feasibility pilot with a single intervention arm, an education control arm, a usual care control arm, and an interview only arm. The intervention arm includes participation in the melodica training program and education about pulmonary health. The education control arm includes pulmonary health education only. The interview only arm includes participation in a semi-structured interview about facilitators and barriers to participation.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Melodica Intervention (Experimental): An 8-week group intervention including twice-weekly sessions. Each session will last one hour in duration with approximately 20 minutes for instruction, 30 minutes in group music-making, and 10 minutes allocated for educational information about COPD, tobacco cessation, and pulmonary rehabilitation.
  Interventions: Behavioral: Melodica Intervention
- Education Control (Active Comparator): A single 90-120 minute education session including the same educational information about COPD, tobacco cessation, and pulmonary rehabilitation provided to the melodica intervention group.
  Interventions: Behavioral: Pulmonary Health Education
- Usual Care Control (No Intervention): Usual care at Richard L. Roudebush VA Medical Center.
- Interview Only (No Intervention): Semi-structured interviews will be conducted with Veterans who meet eligibility criteria, but who do not agree to participate in the intervention, to identify potential barriers to participation

INTERVENTIONS:
Behavioral: Melodica Intervention — The melodica program will include education about pursed lip breathing, instruction in the melodica instrument, and participation in a melodica training group which meets twice-weekly for an 8-week period. Each session will include musical instruction, group music-making, and education about COPD and related health topics.
  Other Names: Melodica Training Program
  Arms: Melodica Intervention
Behavioral: Pulmonary Health Education — A single session including education about COPD and related health topics.
  Arms: Education Control

SUMMARY:
This project seeks to pilot-test the feasibility of using a melodica training program to teach pursed lip breathing for Veterans with chronic obstructive pulmonary disease (COPD) with moderate to severe dyspnea (shortness of breath). Dyspnea occurs commonly among COPD patients and can limit activities of daily living. Pursed lip breathing is a strategy that can improve dyspnea and exercise capacity among COPD patients. The melodica is a musical instrument that looks like a keyboard with a mouthpiece on the side. The melodica is played by exhaling through the mouthpiece while pressing the keys. The MELODY pilot project protocol has been grounded on concepts from occupational therapy; specifically, providing participants with a meaningful new activity that is enjoyable, that can be provided across a spectrum of skill levels, that can provide participants with a new sense of self, and that can improve health outcomes (i.e., dyspnea and exercise endurance).

DETAILED DESCRIPTION:
SPECIFIC AIMS:

Primary Aim 1: Evaluate the safety of a melodica training program to teach pursed lip breathing among Veterans with COPD with moderate to severe dyspnea. We hypothesize that a melodica training program can be safely implemented among COPD patients with severe dyspnea.

Primary Aim 2: Evaluate the feasibility of implementing a melodica training program to teach pursed lip breathing among Veterans with COPD with dyspnea. We hypothesize that it will be feasible to implement a melodica training program to teach pursed lip breathing among Veterans with COPD and dyspnea; specifically that enrolled participants will attend >50% of sessions. We also hypothesize that transportation to the VA Medical Center to attend sessions will be identified as a significant barrier to participation.

Secondary Aim: Collect pilot-efficacy data of a melodica training program to teach pursed lip breathing among Veterans with COPD and dyspnea. The objective is to understand whether melodica training improves dyspnea both in the short-term and in the longer-term over the course of the 8-week training program. We hypothesize that a melodica training program will reduce dyspnea by 30% in the short-term and 10% in the long-term. We also hypothesize that intervention participants will show gains in the secondary efficacy outcome measures of exercise endurance, pulmonary function, entering pulmonary rehabilitation, quality of life, patient global impression of change, and anxiety relative to controls.

RANDOMIZATION AND INTERVENTION:

Randomization:

Participants will be randomized in a 1:1:1 ratio to the intervention group (N=50), usual care control group (N=50), and education control group (N=50) using a block randomization design. We will also seek to identify N=30 Veterans who met the COPD diagnosis and spirometry eligibility criteria but who chose not to participate in the intervention; these Veterans will be invited to participate in a brief interview to identify barriers to participation.

Melodica Program Intervention:

The intervention program will include: education about pursed lip breathing, instruction in the melodica instrument, and participation in a melodica playing group which will meet twice-weekly for a 8-week period. Participants will be given instructional materials for use in practicing the instrument in their homes and encouragement to use pursed lip breathing not only while playing the instrument but also in their activities of daily living. Each session will last one hour in duration with approximately 20 minutes for instruction, 30 minutes in group music-making, and 10 minutes allocated for educational information about COPD, tobacco cessation, and pulmonary rehabilitation.

Education Group:

The patients in the education control group will receive the same educational materials that are provided to the intervention group; however, they will receive them in a single educational session. As described above, the educational materials include information about pursed lip breathing, COPD, medications used to treat COPD, how to use an inhaler, smoking cessation, pulmonary rehabilitation, oxygen therapy, exercise, and travelling with COPD. The materials include handouts as well as links to web pages.

ELIGIBILITY:
Inclusion Criteria:

* spirometry-confirmed COPD defined as a FEV1/FVC <0.7
* moderate or severe dyspnea defined as a grade ≥3 on the ATS Dyspnea scale

Exclusion Criteria:

* visual or hearing impairments
* do not speak English
* do not have an intact airway
* have cognitive impairment
* are unable to make a seal with their mouths
* have a history of at least one hospital admission for congestive heart failure in the prior year
* receiving Hospital-Based Home Care (HBHC) or Telehealth care for COPD management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse Events | Measured at baseline and before and after each of 16 program training sessions (8 week duration).
  We will describe the frequency with which patients reported any adverse events they experienced as a consequence of participation in the program as well as specify the types of adverse events.
Safety: Dyspnea Visual Analog Line | Baseline, before and after each training session (16 sessions over 8 weeks)
  We will measure dyspnea with a visual-analog line (100mm line with anchors at 0=no dyspnea, 100=severe dyspnea)

SECONDARY OUTCOMES:
Feasibility: Program Participation | Measured at baseline
  Feasibility will be measured in terms of the proportion of eligible Veterans who agree to participate
Feasibility: Attendance | Measured at every intervention session (total of 16 sessions over 8 weeks)
  Feasibility will be measured in terms of the proportion of sessions that enrolled participants attend

OTHER OUTCOMES:
Pilot-Efficacy: Dyspnea Visual Analog Line | Baseline, before and after each intervention sessions (16 sessionis over 8 weeks).
  We will measure dyspnea with a visual-analog line (100mm line with anchors at 0=no dyspnea, 100=severe dyspnea)
Secondary Efficacy: Quality of Life (SF-20) | Measured at baseline, 4-weeks, 8-weeks
  We will assess quality of life based on the 20-item Short Form Health Survey (SF-20)
Secondary Efficacy: Exercise Endurance (6-Minute Walk) | Measured at baseline, 4-weeks, 8-weeks
  We will assess exercise endurance measured by the 6-Minute Walk Test (6MWT).

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M Bravata, MD, Principal Investigator — VA Quality Enhancement Research Initiative
Locations (1):
- Veteran Health Indiana, Richard L. Roudebush VA Medical Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McGrath M, Smith J, Rattray NA, Lillie A, Crow S, Myers LJ, Myers J, Perkins AJ, Wasmuth S, Burns DS, Cheatham AJ, Patel H, Bravata DM. Teaching pursed-lip breathing through music: MELodica Orchestra for DYspnea (MELODY) trial rationale and protocol. Arts Health. 2022 Feb;14(1):49-65. doi: 10.1080/17533015.2020.1827277. Epub 2020 Oct 16. PMID 33064621